CLINICAL TRIAL: NCT06906848
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Effects of Cognizin ® Citicoline on Cognitive Performance in Generally Healthy Adults
Brief Title: Evaluate the Effects of Citicoline on Cognitive Performance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirin Holdings Company, Limited (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: K05-24-01-T0060
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Cognitive Performance
Keywords: Citicoline; Cognitive; cognitive performance

STUDY DESIGN:
Intervention Model Description: There are 2 study groups, including one test product (TP) group and one placebo (PL) group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The placebo will match the TP in physical and visual appearance and packaging and each participant's study product assignments will be associated with a unique code to prevent premature unblinding. Planned unblinding will occur following database lock, definition of study populations, and a blinded statistical analysis Delegated unblinded site personnel will be responsible for study product accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records) throughout the course of the study. The investigator will have oversight in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Active ingredients: none
  Interventions: Dietary Supplement: Placebo
- Cognizin® (Active Comparator): Active ingredients: Citicoline
  Interventions: Dietary Supplement: Cognizin®

INTERVENTIONS:
Dietary Supplement: Placebo — Oral
  Arms: Placebo
Dietary Supplement: Cognizin® — Oral
  Other Names: Citicoline supplement
  Arms: Cognizin®

SUMMARY:
Cognizin is a patented form of citicoline, a natural compound of the brain tissue.

It is believed that Cognizin can support brain function by boosting brain energy and protecting brain cells. Research suggests that Cognizin can improve different aspects of brain function and affects cognitive performance in healthy adults.

DETAILED DESCRIPTION:
This study is a prospective, randomized, placebo-controlled, double-blind trial designed to assess the effects of Cognizin on cognitive performance in healthy young adults.

Participants will be randomized in a 1:1 ratio to either the test product (TP) or placebo (PL). During the study, participants cognitive performance will be assessed using the Psychomotor Vigilance Test (PVT) at baseline and after 12 weeks.

Safety assessments will be conducted throughout the study.

Note: The Unique Protocol ID K05-24-01-T0060 was unintentionally combined with another Unique Protocol ID, Bio-2104. As a result, the first protocol record for K05-24-01-T0060 was released in September 2024, prior to participant recruitment and randomization. The study start date was November 2024.

This explanation has been added per PRS instructions to ensure compliance and maintain data integrity in alignment with the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females who are 18-35 years of age (inclusive) at screening.
2. Body mass index (BMI) between 18.0 to 34.9 kg/m2 (inclusive).
3. In good general health and are able to swallow capsules.
4. Participants agree to maintain their usual caffeine consumption habits.
5. Participants who have habitually eaten breakfast for at least 1 month before screening, and agree to eat breakfast daily, and take study product with this meal when applicable as instructed, for the duration of the study.
6. MMSE score >24 at screening.
7. Naïve to oral cannabis or hemp, or light user of oral cannabis or hemp products (not more than 2 times per month on average).
8. Willing and able to agree to the requirements of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study- related procedures.

Exclusion Criteria:

1. Females who are lactating, pregnant or planning to become pregnant during the study.
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
3. Are receiving treatments, or have been hospitalized in the last 12 months, for psychiatric disorders and/or brain-related medical conditions.
4. Participants who have habitually used any nicotine-containing products in the past 6 months before screening.
5. Individuals with any pre-existing neuromuscular disorder, physical disability, or injury.
6. Have inadequate sleep schedule defined as an average of less than 6 hours per night.
7. Have Type I diabetes, uncontrolled Type II diabetes, uncontrolled high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or uncontrolled thyroid disease
8. Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised.
9. Currently have cancer or have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) with recovery occurred at least 5 years before the screening visit.
10. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing and digestion.
11. Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product.
12. Reports a clinically significant illness during the 28 days before the first dose of study product.
13. Major surgery in 3 months prior to screening or planned major surgery during the study.
14. Currently consumes more than two (2) standard alcoholic beverages per day on average for the two weeks prior to screening.
15. Have a history of alcohol or substance abuse in the 12 months prior to screening
16. Current enrolment or past participation in another study with any product(s) with at least one active ingredient within 28 days before first dose of study product or longer.
17. Any other medical condition/situation or use of medications/ supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of the Test Product (TP) on cognitive performance compared to a placebo after 12 weeks using the Psychomotor Vigilance Test (PVT) | 12 weeks

SECONDARY OUTCOMES:
To evaluate the effect of the TP on attention control to a placebo after 12 weeks using the Stroop squared task, Flanker squared task and Simon squared task. | 12 weeks
To evaluate the effect of the TP on motor speed to a placebo after 12 weeks by using the Finger-Tapping test. | 12 weeks

OTHER OUTCOMES:
To assess the safety and tolerability of the TP in healthy participants: Reports of Adverse Events To determine number of participants with adverse events. | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Koichiro Murashima, Study Chair — Kirin Holding Company Ltd. - Institute of Health Sciences
Locations (1):
- Apex Trials, Guelph, Ontario - on, Canada

IPD SHARING:
Plan to Share IPD: No